CLINICAL TRIAL: NCT05913245
Title: Impact of the Preoperative Carbohydrate Loading for Enhancing Recovery After Radical Cystectomy: a Randomized Controlled Trial.
Brief Title: Preoperative Carbohydrate Loading for Enhancing Recovery After Radical Cystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Principal Investigator, Daniel López-Herrera Rodriguez, PhD, Fundación Pública Andaluza para la gestión de la Investigación en Sevilla
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1738-N-22
Record Dates: First submitted 2023-05-30; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Anesthesia; Urologic Cancer; Surgery
Keywords: cystectomy; fasting; preoperative carbohydrate treatment
MeSH Terms: conditions — Urologic Neoplasms; Fasting | interventions — Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fasting arm (No Intervention): Patients included in the fasting arm will not drink or eat anything after the dinner of the night before the surgery.
- Water arm (Active Comparator): Patients included in the water intake arm will drink the same amount of mililiters than the carbohydrate loading drink.
  Interventions: Other: Water
- Carbohydrate loading arm (Experimental): Patients included in the intake arm of carbohydrate loading treatment should take 400ml the night before the intervention and 200ml the two hours before the intervention.
  The hydrocarbonate drink provided will be Sugarmix (Maltodextrin 12.5%).
  Interventions: Dietary Supplement: Maltodextrin 12.5%

INTERVENTIONS:
Dietary Supplement: Maltodextrin 12.5% — Preoperative Maltodextrin 12.5%
  Arms: Carbohydrate loading arm
Other: Water — Preoperative water
  Arms: Water arm

SUMMARY:
In recent years, the world of anesthesiology is questioning one of its great dogmas: Are so many hours of strict fasting necessary in patients who are candidates for elective surgeries? The main objective of our clinical trial will be demonstrate whether preoperative oral loading with hydrocarbonate beverages reduces the time of return of intestinal function in the postoperative period compared to water administration and strict fasting in patients undergoing elective radical cystectomy.

DETAILED DESCRIPTION:
Many anaesthesiology societies now recommend intake of clear fluids (water, tea or coffee without milk, juices without pulp) up to two hours before induction of anaesthesia for most patients undergoing elective surgery. This change the traditional practice of overnight fasting, while reducing thirst in the hours before surgery and seems to attenuate the response to the stress that results from a major operation, such as activation of endocrine and inflammatory systems which leads to tissue catabolism and insulin resistance. Among all the complications, one of the most frequent in patients undergoing mayor surgeries is undoubtedly paralytic ileus. The Enhanced Recovery After Surgery (ERAS) guidelines emphasize the importance of preventing this event. To prevent ileus, prokinetic agents such as metoclopramide are used, which although it has not been shown to shorten the period until the first flatulence or the first peristaltic movement, decrease nausea and vomiting. Chewing gum is another measure that is carried out, since it stimulates peristalsis and this measure if it had significant effects in time until first flatulence and in time until first peristaltic movement. In recent years there has been a great change in the perioperative management of patients who will undergo a radical cystectomy. The weight of traditional perioperative care has been an important barrier to the implementation of Fast Track (FT) protocols, since it is difficult to change a therapeutic strategy that has been carried out for decades. The positive results obtained in colorectal surgery led to Fast Track being implemented in other types of surgery similar to colorectal surgery such as radical cystectomy. Although there is apparently widespread enthusiasm for the implementation of Fast Track protocols, evidence of the use of this type of protocols in cystectomy is not robust, numerous studies claim that there is a big difference between the application of FT and the application of traditional measures in terms of length of hospital stay or complications. Because of this, more large-volume randomized experimental studies of patients are needed. This randomized double blind placebo-controlled trial of preoperative oral carbohydrate (CHO) treatment in patients undergoing elective radical cystectomy will investigate whether this treatment reduced the time of return of intestinal function. Secondary outcomes will be the incidence of infection of surgical wounds, the incidence of postoperative complications, the length of hospital stay and early postoperative fatigue in the three groups of patients undergoing this type of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Patients older than 18 years old proposed for radical cystectomy.

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) classification grade: IV
* Renal failure (creatinine levels above 3 mg/dL or dialysis)
* Liver failure (Child-Pugh B or higher)
* Gastroesophageal reflux disease.
* Gastrointestinal obstruction.
* Ongoing treatment with corticosteroids.
* Previous infections within the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Insulin resistance | 1 Day of surgery
  Determinate the insulin resistance measured by the homeostatic model assessment (HOMA) index.

SECONDARY OUTCOMES:
To determine the recovery time of intestinal activity by measuring time to first bowel movement. | 1 week
  Bowel movement
To compare and determine whether there are differences between the incidence of infection of surgical wounds, the incidence of postoperative complications and the length of hospital stay in the three groups of patients undergoing this type of surgery. | Up to 30 days
  Complications
Insulin resistance | Postoperative day #1
  Determinate the insulin resistance measured by the homeostatic model assessment

CONTACTS AND LOCATIONS:
Overall Officials: Clara Rosso, PhD, Study Chair — Fundación Pública Andaluza para la gestión de la Investigación en Sevilla
Locations (1):
- Fundación Pública Andaluza para la Gestión de Investigación de Salud en Sevilla, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial. Study Protocol, Statistical Analysis Plan, Inform Consent Form, Clinical
  Study Report and Analytic Code will also be available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication and with no end date.
Access Criteria: Researchers who provide a methodologically sound proposal to achieve aims in the approved proposal.